CLINICAL TRIAL: NCT05276778
Title: Diabetic Retinopathy Screenings in General Practice for People With Type 2 Diabetes
Brief Title: Diabetic Retinopathy Screening in General Practice
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Malene Krogh, Ph.D. student, Aalborg University
Other Study IDs: mKrogh
Record Dates: First submitted 2022-02-28; First posted 2022-03-11 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2023-01

CONDITIONS: Diabetic Retinopathy; Type2 Diabetes
Keywords: Artificial Intelligence; Diabetic Retinopathy Screening; General practice; Primary care; Type 2 diabetes
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- People with type 2 diabetes: People diagnosed with type 2 diabetes age 18-70
  Interventions: Diagnostic Test: Diabetic Retinopathy Screening

INTERVENTIONS:
Diagnostic Test: Diabetic Retinopathy Screening — Screenings are performed in the diabetes consultation in general practice

SUMMARY:
Diabetic Retinopathy is a microvascular eye complication of diabetes, which can go unnoticed until permanent vision damage has occurred - in worst-case blindness. Timely retinopathy screenings reduce the risk of sight loss since the disease can be treated if detected in time. For people with type 2 diabetes, retinopathy screenings are typically performed by specialist at private ophthalmologists' practices, and individualized screening intervals based on retinopathy level and diabetes regulation are recommended. Unfortunately, 26% of people with type 2 diabetes do not follow their screening interval, and the attendance is too low compared to the national standard of minimum 90% of patients with diabetes who ought to follow the screening program. Consequently, actions must be taken to improve screening attendance in Denmark.

The aim of this study is to investigate patients' acceptance of diabetic retinopathy screenings in general practice. Patients' acceptance is explored through a questionnaire developed for the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* Understands Danish
* Age between 18-70

Exclusion Criteria:

* Blindness
* Cannot partake in second screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients diagnosed with type 2 diabetes treated in general practice within the Region of North Jutland. We are excluding patients above the age of 70 as patients at this age diagnosed with diabetes have a higher risk of developing other eye diseases, such as glaucoma or cataracts, so the general practitioners would still have to advice this patient group to schedule consultations at an ophthalmologist even though they have no sign of retinopathy.
  Patients who participate in the project must fulfill all inclusion criteria and cannot fulfill any exclusion criteria listed below.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Patients' acceptance of diabetic retinopathy screenings in general practice | 1 day (the questionnarie is fufilled one time after the retinopaty screening in general practice)
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Malene Krogh, Principal Investigator — Aalborg University
Locations (1):
- Malene Krogh, Aalborg, DK, Denmark

IPD SHARING:
Plan to Share IPD: Undecided